CLINICAL TRIAL: NCT04072978
Title: Anterior Chamber Versus Scleral Fixated Intraocular Lens: Long-term Vision and Safety Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Kertes, Ophthalmologist - Retina Specialist, Sunnybrook Health Sciences Centre
Other Study IDs: 00046460
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Corneal Endothelial Cell Loss; Secondary Intraocular Lens
MeSH Terms: conditions — Corneal Endothelial Cell Loss | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Intraocular lens implantation: AC IOL: Patients who are scheduled to undergo AC IOL (anterior chamber intraocular lens) implantation for any of the following indications:
  * primary or secondary aphakia
  * primary or secondary lens subluxation or dislocation
  Interventions: Device: Intraocular lens implantation
- Intraocular lens implantation: SF IOL: Patients who are scheduled to undergo SF IOL (scleral fixated intraocular lens) implantation for any of the following indications:
  * primary or secondary aphakia
  * primary or secondary lens subluxation or dislocation
  Interventions: Device: Intraocular lens implantation

INTERVENTIONS:
Device: Intraocular lens implantation — Implantation of an intraocular lens using either an anterior chamber IOL or a scleral fixated IOL using the modified Yamane technique.
  Other Names: IOL implantation

SUMMARY:
This is a prospective comparative non-randomized cohort study to understand the long-term vision outcomes, safety, and stability of anterior chamber intraocular lenses (AC IOLs) vs. scleral-fixated intraocular lenses (SF IOLs).

DETAILED DESCRIPTION:
On the pre-operative visit, specular microscopy, biometry, applanation tonometry and ocular coherence tomography (OCT) will be performed. The patient will then undergo treatment as per surgeon's discussion/ decision with the patient for implantation of an AC-IOL or SF-IOL. Participation in the study will not impact the management plan in any way. Specular microscopy will be performed wit the CellChek XL (Konan Medical, Irvine, CA). Biometry will be performed with the IOLMASTER (Carl Ziess Meditec, Jena, Germany), and anterior segment and macular OCT will be performed with the Cirrus-HD OCT (Carl Zeiss Metidec, Jena, Germany). EC count, OCT (macula and anterior segment) and specular microscopy will be performed at baseline, week 1, month 1, month 6, 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing AC IOL or SF IOL implantation for any reason (including but not limited to aphakia, posterior capsular rupture, primary or secondary lens dislocation/ subluxation or IOL exchange).
2. Patients on whom imaging (specular microscopy, biometry and OCT) can be performed without delaying their treatment (i.e. based on availability of operator).
3. Decision makers able to provide informed consent.

Exclusion Criteria:

1. Inability to obtain adequate imaging, in the form of specular microscopy and OCT data at baseline.
2. Patients unable to attend follow-up visits.
3. Patients who have had a corneal transplant prior to secondary IOL implantation.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are planned to undergo surgical implantation of an anterior chamber intraocular lens or a scleral-fixated IOL who present to the study investigators as part of the vitreoretinal surgery team at Sunnybrook Hospital or the Toronto Western Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell loss | Pre-operative (baseline) and 24 weeks post-operatively.
  Change in endothelial cell count from baseline compared to 24 months post-operatively.

SECONDARY OUTCOMES:
Corrected distance visual acuity (CDVA) | Pre-operative (baseline), week 1, months 1, 6, 12 and 24 post-operatively.
  CDVA will be measured using a standardized Early Treatment Diabetic Retinopathy Study (ETDRS) chart

OTHER OUTCOMES:
Secondary adverse events (SAE's) | Pre-operative (baseline), week 1, months 1, 6, 12 and 24 post-operatively.
  Occurrence of cystoid macular edema (CME), retinal detachment, UGH syndrome, vitreous or choroidal hemorrhage, lens subluxation/ dislocation, glaucoma, uveitis, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kertes, MD, Principal Investigator — Sunnybrook Hospital
Locations (1):
- Sunnybrook Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan TC, Lam JK, Jhanji V, Li EY. Comparison of outcomes of primary anterior chamber versus secondary scleral-fixated intraocular lens implantation in complicated cataract surgeries. Am J Ophthalmol. 2015 Feb;159(2):221-6.e2. doi: 10.1016/j.ajo.2014.10.016. Epub 2014 Oct 22. PMID 25448990
- [Background] Krysik K, Dobrowolski D, Wroblewska-Czajka E, Lyssek-Boron A, Wylegala E. Comparison of the Techniques of Secondary Intraocular Lens Implantation after Penetrating Keratoplasty. J Ophthalmol. 2018 Sep 12;2018:3271017. doi: 10.1155/2018/3271017. eCollection 2018. PMID 30298105
- [Background] Kwong YY, Yuen HK, Lam RF, Lee VY, Rao SK, Lam DS. Comparison of outcomes of primary scleral-fixated versus primary anterior chamber intraocular lens implantation in complicated cataract surgeries. Ophthalmology. 2007 Jan;114(1):80-5. doi: 10.1016/j.ophtha.2005.11.024. Epub 2006 Oct 27. PMID 17070590
- [Background] Negretti GS, Lai M, Petrou P, Walker R, Charteris D. Anterior chamber lens implantation in vitrectomised eyes. Eye (Lond). 2018 Mar;32(3):597-601. doi: 10.1038/eye.2017.261. Epub 2017 Dec 8. PMID 29219957
- [Background] Yamane S, Sato S, Maruyama-Inoue M, Kadonosono K. Flanged Intrascleral Intraocular Lens Fixation with Double-Needle Technique. Ophthalmology. 2017 Aug;124(8):1136-1142. doi: 10.1016/j.ophtha.2017.03.036. Epub 2017 Apr 27. PMID 28457613
- [Background] Brunin G, Sajjad A, Kim EJ, Montes de Oca I, Weikert MP, Wang L, Koch DD, Al-Mohtaseb Z. Secondary intraocular lens implantation: Complication rates, visual acuity, and refractive outcomes. J Cataract Refract Surg. 2017 Mar;43(3):369-376. doi: 10.1016/j.jcrs.2016.12.024. PMID 28410720